CLINICAL TRIAL: NCT01960348
Title: APOLLO: A Phase 3 Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Patisiran (ALN-TTR02) in Transthyretin (TTR)-Mediated Polyneuropathy (Familial Amyloidotic Polyneuropathy-FAP)
Brief Title: APOLLO: The Study of an Investigational Drug, Patisiran (ALN-TTR02), for the Treatment of Transthyretin (TTR)-Mediated Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-TTR02-004; 2013-002987-17 (EudraCT Number)
Expanded Access: NCT02939820 (Approved for marketing)
Record Dates: First submitted 2013-10-09; First posted 2013-10-10 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2018-11

CONDITIONS: TTR-mediated Amyloidosis; Amyloidosis, Hereditary; Amyloid Neuropathies, Familial; Familial Amyloid Polyneuropathies; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related
Keywords: RNAi therapeutic; FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — patisiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patisiran (ALN-TTR02) (Active Comparator)
  Interventions: Drug: patisiran (ALN-TTR02)
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: patisiran (ALN-TTR02) — administered by intravenous (IV) infusion
  Arms: patisiran (ALN-TTR02)
Drug: Sterile Normal Saline (0.9% NaCl) — administered by intravenous (IV) infusion
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of patisiran (ALN-TTR02) in patients with transthyretin (TTR) mediated amyloidosis. An open-label, single-arm, long-term follow-up extension study NCT02510261 (ALN-TTR02-006) was initiated to provide participants who completed this study with continued patisiran-LNP (lipid nanoparticle) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 85 years of age (inclusive);
* Have a diagnosis of FAP
* Neuropathy Impairment Score requirement of 5-130
* Meet Karnofsky performance status requirements
* Have adequate complete blood counts and liver function tests
* Have adequate cardiac function
* Have negative serology for hepatitis B virus (HBV) and hepatitis C virus (HCV)

Exclusion Criteria:

* Had a prior liver transplant or is planned to undergo liver transplant during the study period;
* Has untreated hypo- or hyperthyroidism;
* Has known human immunodeficiency virus (HIV) infection;
* Had a malignancy within 2 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated;
* Recently received an investigational agent or device
* Is currently taking diflunisal, tafamidis, doxycycline, or tauroursodeoxycholic acid

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, Study Director — Alnylam Pharmaceuticals
Locations (49):
- United States (12):
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Portland, Oregon
- Clinical Trial Site, Buenos Aires, Argentina
- Clinical Trial Site, Westmead, Australia
- Brazil (3):
  - Clinical Trial Site, Ribeirão Preto
  - Clinical Trial Site, Rio de Janeiro
  - Clinical Trial Site, São Paulo
- Clinical Trial Site, Sofia, Bulgaria
- Clinical Trial Site, Vancouver, British Columbia, Canada
- Clinical Trial Site, Nicosia, Cyprus
- France (5):
  - Clinical Trial Site, Bourdeaux
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Marseille
- Germany (3):
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Münster
  - Clinical Trial Site, Regensburg
- Italy (3):
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Rome
  - Clinical Trial Site, Sicily
- Japan (3):
  - Clinical Trial Site, Matsumoto, Nagano
  - Clinical Trial Site, Aichi
  - Clinical Trial Site, Kumamoto
- Clinical Trial Site, Kuala Lumpur, Malaysia
- Clinical Trial Site, Mexico City, Mexico
- Clinical Trial Site, Groningen, Netherlands
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Clinical Trial Site, Seoul, South Korea
- Spain (4):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Huelva
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Palma de Mallorca
- Clinical Trial Site, Umeå, Sweden
- Taiwan (2):
  - Clinical Trial Site, Taipai
  - Clinical Trial Site, Taipei
- Clinical Trial Site, Istanbul, Turkey (Türkiye)
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Lin KP, Yang CC, Lee YC, Lee MJ, Vest J, Sweetser MT, White MT, Badri P, Hsieh ST, Chao CC. Patisiran, an RNAi therapeutic for hereditary transthyretin-mediated amyloidosis: Sub-analysis in Taiwanese patients from the APOLLO study. J Formos Med Assoc. 2024 Sep;123(9):975-984. doi: 10.1016/j.jfma.2024.03.008. Epub 2024 Mar 27. PMID 38548524
- [Derived] Quan D, Obici L, Berk JL, Ando Y, Aldinc E, White MT, Adams D. Impact of baseline polyneuropathy severity on patisiran treatment outcomes in the APOLLO trial. Amyloid. 2023 Mar;30(1):49-58. doi: 10.1080/13506129.2022.2118043. Epub 2022 Sep 18. PMID 36120830
- [Derived] Zhang X, Goel V, Attarwala H, Sweetser MT, Clausen VA, Robbie GJ. Patisiran Pharmacokinetics, Pharmacodynamics, and Exposure-Response Analyses in the Phase 3 APOLLO Trial in Patients With Hereditary Transthyretin-Mediated (hATTR) Amyloidosis. J Clin Pharmacol. 2020 Jan;60(1):37-49. doi: 10.1002/jcph.1480. Epub 2019 Jul 19. PMID 31322739
- [Derived] Minamisawa M, Claggett B, Adams D, Kristen AV, Merlini G, Slama MS, Dispenzieri A, Shah AM, Falk RH, Karsten V, Sweetser MT, Chen J, Riese R, Vest J, Solomon SD. Association of Patisiran, an RNA Interference Therapeutic, With Regional Left Ventricular Myocardial Strain in Hereditary Transthyretin Amyloidosis: The APOLLO Study. JAMA Cardiol. 2019 May 1;4(5):466-472. doi: 10.1001/jamacardio.2019.0849. PMID 30878017
- [Derived] Solomon SD, Adams D, Kristen A, Grogan M, Gonzalez-Duarte A, Maurer MS, Merlini G, Damy T, Slama MS, Brannagan TH 3rd, Dispenzieri A, Berk JL, Shah AM, Garg P, Vaishnaw A, Karsten V, Chen J, Gollob J, Vest J, Suhr O. Effects of Patisiran, an RNA Interference Therapeutic, on Cardiac Parameters in Patients With Hereditary Transthyretin-Mediated Amyloidosis. Circulation. 2019 Jan 22;139(4):431-443. doi: 10.1161/CIRCULATIONAHA.118.035831. PMID 30586695
- [Derived] Adams D, Gonzalez-Duarte A, O'Riordan WD, Yang CC, Ueda M, Kristen AV, Tournev I, Schmidt HH, Coelho T, Berk JL, Lin KP, Vita G, Attarian S, Plante-Bordeneuve V, Mezei MM, Campistol JM, Buades J, Brannagan TH 3rd, Kim BJ, Oh J, Parman Y, Sekijima Y, Hawkins PN, Solomon SD, Polydefkis M, Dyck PJ, Gandhi PJ, Goyal S, Chen J, Strahs AL, Nochur SV, Sweetser MT, Garg PP, Vaishnaw AK, Gollob JA, Suhr OB. Patisiran, an RNAi Therapeutic, for Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):11-21. doi: 10.1056/NEJMoa1716153. PMID 29972753
- [Derived] Adams D, Suhr OB, Dyck PJ, Litchy WJ, Leahy RG, Chen J, Gollob J, Coelho T. Trial design and rationale for APOLLO, a Phase 3, placebo-controlled study of patisiran in patients with hereditary ATTR amyloidosis with polyneuropathy. BMC Neurol. 2017 Sep 11;17(1):181. doi: 10.1186/s12883-017-0948-5. PMID 28893208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 225 patients with hereditary transthyretin (hATTR) amyloidosis were enrolled and randomized in the study.
Groups:
- Patisiran (ALN-TTR02): All patients who received at least 1 dose of patisiran (ALN-TTR02)
- Placebo: All patients who received at least 1 dose of placebo
Period: Overall Study
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Started | 148 | 77
Completed (Participants who completed this study could enter the extension study NCT02510261 (ALN-TTR02-006)) | 138 | 55
Not Completed | 10 | 22
Not completed — Adverse event, not serious | 2 | 2
Not completed — Adverse event, serious fatal | 6 | 5
Not completed — Adverse event, serious non-fatal | 0 | 3
Not completed — Withdrawal by Subject | 1 | 11
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patisiran (ALN-TTR02) | Placebo | Total
Number analyzed (Participants) | 148 | 77 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.96) | 62.2 (10.76) | 60.5 (11.61)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 86 | 44 | 130
  65-74 years | 53 | 24 | 77
  ≥75 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 19 | 58
  Male | 109 | 58 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 130 | 65 | 195
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 25 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 113 | 50 | 163
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Baseline NIS [Count of Participants; unit: Participants] — The Neuropathy Impairment Score is an assessment of motor weakness (NIS-W), sensation (NIS-S) and reflexes (NIS-R) scored based on physical exam findings.
  NIS-W is a measure of motor strength, comprised of cranial nerve and both upper and lower limb motor assessments. The minimum and maximum values are 0 and 192, respectively. A higher score indicates a worse outcome.
  Participants
    NIS <50 | 62 | 35 | 97
    NIS ≥50 | 86 | 42 | 128
Genotype Class [Count of Participants; unit: Participants] — Transthyretin (TTR) genotype class, collected at baseline
  Participants
    Early onset V30M (<50 years of age at onset) | 13 | 10 | 23
    All other mutations (including late onset V30M) | 135 | 67 | 202
Previous Tetramer Stabilizer Use [Count of Participants; unit: Participants] — Prior use of tafamidis meglumine or diflunisal
  Participants
    Yes | 78 | 41 | 119
    No | 70 | 36 | 106
Baseline mNIS+7 [Mean (Standard Deviation); unit: Points] — The mNIS+7 is a composite score that quantitates motor, sensory, and autonomic neurologic impairment due to injury of large and small nerves. The minimum and maximum values are 0 and 304, respectively. A higher score indicates a worse outcome.
  Points | 80.93 (41.507) | 74.61 (37.041) | 78.77 (40.064)

OUTCOME MEASURES:

1. Primary Outcome: Modified Neuropathy Impairment Score +7 (mNIS+7)
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in mNIS+7 at 18 months. The mNIS+7 is a composite score that quantitates motor, sensory, and autonomic neurologic impairment due to injury of large and small nerves. The minimum and maximum values are 0 and 304, respectively. A higher score indicates a worse outcome.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month mNIS+7 assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 137 | 51
score on a scale | -6.03 (1.739) | 27.96 (2.602)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in mNIS+7. The model includes baseline mNIS+7 score as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=9.262E-24; Least Squares Mean Difference = -33.99, 95% CI 2-sided [-39.86 to -28.13], Standard Error of Mean 2.974

2. Secondary Outcome: Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QoL-DN) Questionnaire
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in Norfolk QoL-DN at 18 months. The Norfolk QoL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy - small fiber, large fiber, and autonomic nerve function. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month Norfolk QoL-DN assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 136 | 48
score on a scale | -6.7 (1.77) | 14.4 (2.73)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in Norfolk QOL-DN total score. The model includes baseline Norfolk QOL-DN score as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline NIS, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=1.103E-10; Least Squares Mean Difference = -21.1, 95% CI 2-sided [-27.2 to -15.0], Standard Error of Mean 3.10

3. Secondary Outcome: Neurological Impairment Score-Weakness (NIS-W) Score
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in NIS-W at 18 months. NIS-W is a measure of motor strength, comprised of cranial nerve and both upper and lower limb motor assessments. The minimum and maximum values are 0 and 192, respectively. A higher score indicates a worse outcome.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month NIS-W assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 137 | 51
score on a scale | 0.05 (1.306) | 17.93 (1.959)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in NIS-W. The model includes baseline NIS-W score as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=1.404E-13; Least Squares Mean Difference = -17.87, 95% CI 2-sided [-22.32 to -13.43], Standard Error of Mean 2.254

4. Secondary Outcome: Rasch-built Overall Disability Scale (R-ODS) Score
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in R-ODS score at 18 months. The R-ODS is comprised of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients. The minimum and maximum values are 0 and 48, respectively. A higher score indicates a better outcome.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and either the 18-month R-ODS assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 138 | 54
score on a scale | 0.0 (0.59) | -8.9 (0.88)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in R-ODS value. The model includes baseline R-ODS score as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline NIS, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=4.066E-16; Least Squares Mean Difference = 9.0, 95% CI 2-sided [7.0 to 10.9], Standard Error of Mean 1.01

5. Secondary Outcome: Timed 10-meter Walk Test (10-MWT, Gait Speed)
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in 10-MWT at 18 months. Ability to ambulate (gait speed) was assessed through the 10-meter walk test (10-MWT). The walk had to be completed without assistance from another person; ambulatory aids such as canes and walkers were permitted.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month 10-MWT assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 138 | 55
m/sec | 0.077 (0.0242) | -0.235 (0.0358)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in 10-meter walk test result. The model includes baseline 10-meter walk test result as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline NIS, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=1.875E-12; Least Squares Mean Difference = 0.311, 95% CI 2-sided [0.230 to 0.393], Standard Error of Mean 0.0415

6. Secondary Outcome: Modified Body Mass Index (mBMI)
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in mBMI at 18 months. The nutritional status of patients was evaluated using the mBMI; calculated as the product of BMI (weight in kilograms divided by the square of height in meters) and serum albumin (g/L).
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month mBMI assessments and did not experience any major protocol deviations that may have impacted the results..
Measure: Least Squares Mean (Standard Error); unit: kg/m^2 × albumin g/L
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 133 | 52
kg/m^2 × albumin g/L | -3.7 (9.57) | -119.4 (14.51)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in mBMI. The model includes baseline mBMI as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline NIS, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p < 0.0000001, Mixed-effect Model Repeated Measures — P=8.832E-11; Least Squares Mean Difference = 115.7, 95% CI 2-sided [82.4 to 149.0], Standard Error of Mean 16.91

7. Secondary Outcome: Autonomic Symptoms Questionnaire (Composite Autonomic Symptom Score [COMPASS 31])
Description: The difference between the patisiran (ALN-TTR02) and placebo groups in the change from baseline in COMPASS 31 at 18 months. The COMPASS 31 is a measure of autonomic neuropathy symptoms. The questions evaluated 6 autonomic domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor). The minimum and maximum values are 0 and 100, respectively. A higher score indicates a worse outcome.
Time Frame: 18mo
Population: Per protocol (PP) population: All randomized participants who received at least 1 dose of patisiran-LNP or placebo, completed baseline and the 18-month COMPASS 31 assessments, and did not experience any major protocol deviations that may have impacted the efficacy results.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran (ALN-TTR02) | Placebo
Number analyzed (Participants) | 136 | 53
score on a scale | -5.29 (1.300) | 2.24 (1.940)
Statistical Analysis 1: Comparison: Patisiran (ALN-TTR02) vs Placebo; In the mixed-effect model repeated measures (MMRM) model, the outcome variable is change from baseline in COMPASS-31 total score. The model includes baseline COMPASS-31 score as covariate and fixed effect terms including treatment group, visit, treatment-by-visit interaction, baseline NIS, genotype, age at hATTR symptom onset, previous tetramer stabilizer use and region; Test type: Superiority; p = 0.0008, Mixed-effect Model Repeated Measures; Least Squares Mean Difference = -7.53, 95% CI 2-sided [-11.89 to -3.16], Standard Error of Mean 2.213

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) that occurred from start of study drug administration through End of Study (Day 567), or Follow-up (Day 602) if patient did not enter open-label extension study. AEs for patients with Rapid Disease Progression at Month 9 who stopped dosing were collected through Day 294 (42 days after last dose).
Description: The same event may appear as both an AE and a Serious Adverse Event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Safety population: All participants who received at least 1 dose of patisiran-LNP or placebo. Participants were analyzed according to the treatment received.
Arm/Group | Patisiran (ALN-TTR02) | Placebo
All-Cause Mortality (participants affected / at risk) | 7/148 | 6/77
Serious Adverse Events (participants affected / at risk) | 54/148 | 31/77
Other Adverse Events (participants affected / at risk) | 143/148 | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patisiran (ALN-TTR02) (N=148) | Placebo (N=77)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Syringomyelia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (4)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Device battery issue (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2)
Infected skin ulcer (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug level increased (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 4 (5)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Liver transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patisiran (ALN-TTR02) (N=148) | Placebo (N=77)
Diarrhoea (Gastrointestinal disorders) | 50 (156) | 28 (94)
Oedema peripheral (General disorders) | 43 (68) | 17 (35)
Infusion related reaction (Immune system disorders) | 28 (145) | 7 (79)
Fall (Injury, poisoning and procedural complications) | 25 (47) | 22 (42)
Constipation (Gastrointestinal disorders) | 22 (29) | 12 (17)
Nausea (Gastrointestinal disorders) | 22 (50) | 16 (22)
Dizziness (Nervous system disorders) | 19 (24) | 11 (37)
Urinary tract infection (Infections and infestations) | 19 (40) | 12 (18)
Fatigue (General disorders) | 18 (27) | 8 (18)
Headache (Nervous system disorders) | 16 (25) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 9 (11)
Insomnia (Psychiatric disorders) | 15 (24) | 7 (12)
Nasopharyngitis (Infections and infestations) | 15 (26) | 6 (11)
Asthenia (General disorders) | 14 (25) | 8 (11)
Vomiting (Gastrointestinal disorders) | 14 (20) | 6 (27)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 12 (23) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (18) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 11 (12) | 5 (6)
Influenza (Infections and infestations) | 11 (13) | 4 (4)
Pyrexia (General disorders) | 11 (12) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (9)
Erythema (Skin and subcutaneous tissue disorders) | 10 (51) | 2 (2)
Neuralgia (Nervous system disorders) | 10 (29) | 5 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (12)
Bronchitis (Infections and infestations) | 9 (11) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 0 (0)
Balance disorder (Nervous system disorders) | 8 (10) | 2 (2)
Cataract (Eye disorders) | 8 (10) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 5 (5)
Hypotension (Vascular disorders) | 8 (8) | 5 (9)
Paraesthesia (Nervous system disorders) | 8 (23) | 3 (5)
Vertigo (Ear and labyrinth disorders) | 8 (11) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 7 (7) | 6 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 5 (9)
Haematuria (Renal and urinary disorders) | 6 (9) | 7 (12)
Weight decreased (Investigations) | 6 (6) | 7 (7)
Depression (Psychiatric disorders) | 5 (5) | 5 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (8) | 11 (17)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
Somnolence (Nervous system disorders) | 5 (13) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (5) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 4 (6) | 5 (5)
Peripheral swelling (General disorders) | 4 (6) | 4 (6)
Thermal burn (Injury, poisoning and procedural complications) | 4 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 6 (8)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 8 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 5 (6)
Syncope (Nervous system disorders) | 2 (2) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 1 (3) | 5 (7)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT01960348/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT01960348/SAP_001.pdf